CLINICAL TRIAL: NCT00823615
Title: Comparison of Two New Silicone Hydrogel Multifocal Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-319-C-005 sub 7
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lotrafilcon B / Senofilcon A (Other): Lotrafilcon B, followed by Senofilcon A
  Interventions: Device: Lotrafilcon B multifocal contact lens; Device: Senofilcon A multifocal contact lens
- Senofilcon A / Lotrafilcon B (Other): Senofilcon A, followed by Lotrafilcon B
  Interventions: Device: Lotrafilcon B multifocal contact lens; Device: Senofilcon A multifocal contact lens

INTERVENTIONS:
Device: Lotrafilcon B multifocal contact lens — Silicone hydrogel, soft, multifocal contact lens for daily wear use
Device: Senofilcon A multifocal contact lens — Silicone hydrogel, soft, multifocal contact lens for daily wear use

SUMMARY:
The purpose of this trial is to compare the performance of two multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* At least 35 years of age
* Best-corrected visual acuity of at least 20/40 in each eye.
* Spectacle add between +0.75D and +1.50D (inclusive).
* Able to be fit in available study sphere powers (-0.50 to -5.50D).
* Currently wearing soft contact lenses at least 5 days a week.
* Other protocol inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Eye injury or surgery within twelve weeks immediately prior to enrollment.
* Currently enrolled in an ophthalmic Clinical Trial.
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Previous refractive surgery.
* Astigmatism > 1.00D.
* Currently wearing ACUVUE OASYS for PRESBYOPIA.
* Other protocol inclusion/exclusion criteria may apply.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were enrolled but not dispensed due to failing inclusion criteria. These participants were included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Groups:
- Lotrafilcon B / Senofilcon A: Lotrafilcon B multifocal contact lens worn first, followed by Senofilcon A multifocal contact lens worn second. Both products were worn on a daily-wear basis.
- Senofilcon A / Lotrafilcon B: Senofilcon A multifocal contact lens worn first, followed by Lotrafilcon B multifocal contact lens worn second. Both products were worn on a daily-wear basis.
Period: Period 1
Arm/Group | Lotrafilcon B / Senofilcon A | Senofilcon A / Lotrafilcon B
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Lotrafilcon B / Senofilcon A | Senofilcon A / Lotrafilcon B
Started | 19 | 19
Completed | 16 | 17
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Time/Job Conflict | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed subjects
Arm/Group | Overall
Number analyzed (Participants) | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 47.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Corrected Distance Binocular Visual Measurement in Normal Illumination Reported as Binocular Distance Visual Acuity
Description: Tested while reading charts distant to the subject with both eyes together in normal lighting. This outcome is measured in logMAR units (logarithm of the minimum angle of resolution). A logMAR acuity of 0.0 equates to 20/20 Snellen acuity and is considered normal. Positive logMAR values indicate poorer vision and negative values denote better visual acuity.
Time Frame: After 1 week of wear
Population: Per protocol. Analysis excluded major protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Lotrafilcon B Multifocal Contact Lens; Senofilcon A Multifocal Contact Lens: Silicone hydrogel, soft, multifocal contact lens
Arm/Group | Lotrafilcon B Multifocal Contact Lens | Senofilcon A Multifocal Contact Lens
Number analyzed (Participants) | 33 | 33
LogMAR | -0.08 (0.04) | -0.04 (0.06)

2. Primary Outcome: Corrected Near Binocular Visual Measurement in Normal Illumination Reported as Binocular Near Visual Acuity
Description: Tested while reading charts at 40 cm with both eyes together in normal lighting. This outcome is measured in logMAR units (logarithm of the minimum angle of resolution). A logMAR acuity of 0.0 equates to 20/20 Snellen acuity and is considered normal. Positive logMAR values indicate poorer vision and negative values denote better visual acuity.
Time Frame: After 1 week of wear
Population: Per protocol. Analysis excluded major protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Lotrafilcon B Multifocal Contact Lens | Senofilcon A Multifocal Contact Lens
Number analyzed (Participants) | 33 | 33
LogMAR | 0.05 (0.11) | 0.10 (0.14)

ADVERSE EVENTS:
Time Frame: 9 weeks, duration of the study
Description: 1 week of wear for each intervention
Arm/Group | Lotrafilcon B Multifocal Contact Lens | Senofilcon A Multifocal Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/39 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any pre-clinical and/or clinical data or impressions from this trial.